CLINICAL TRIAL: NCT04259983
Title: Investigation of the Relationship Between Micro and Macrovascular Functions and Exercise Capacity and Respiratory Functions in Children With Cystic Fibrosis of Different Obstruction Severities
Brief Title: Investigation of Relationship Between Vascular Functions, Exercise Capacity, and Respiratory Functions in CF
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Senem Simsek, Principal Investigator, Hacettepe University
Other Study IDs: GO19/1156
Record Dates: First submitted 2020-01-28; First posted 2020-02-07 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Cystic Fibrosis
Keywords: Endothelial Dysfunction; Arterial Stiffness; Exercise Capacity; Respiratory Functions; Children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with CF with normal obstruction severity: In CF children with normal obstruction severity will be subjected to the same maximal exercise test, endothelial dysfunction and arterial stiffness assessments.
  Interventions: Other: Maximal exercise test; Other: Endothelial dysfunction assessment; Other: Arterial stiffness assessment
- Patients with CF with mild obstruction severity: In CF children with mild obstruction severity will be subjected to the same maximal exercise test, endothelial dysfunction and arterial stiffness assessments.
  Interventions: Other: Maximal exercise test; Other: Endothelial dysfunction assessment; Other: Arterial stiffness assessment
- Patients with CF with moderate obstruction severity: In CF children with moderate obstruction severity will be subjected to the same maximal exercise test, endothelial dysfunction and arterial stiffness assessments.
  Interventions: Other: Maximal exercise test; Other: Endothelial dysfunction assessment; Other: Arterial stiffness assessment

INTERVENTIONS:
Other: Maximal exercise test — The maximal exercise test will be performed on an electronically braked bicycle ergometer.
Other: Endothelial dysfunction assessment — Endothelial dysfunction will be determined by blood samples. Blood samples will be collected and analyzed for the responses of ICAM-1, VCAM-1, E-Selectin, VEGF, ET-1.
Other: Arterial stiffness assessment — Arterial stiffness, oscillometric pulse wave velocity (PWV) and augmentation index will be evaluated by recorded brachial pulse waves with automatically with the oscillometric device.

SUMMARY:
In the literature, there is no study that evaluates the endothelial function and arterial stiffness together and investigates its relationship with exercise capacity and respiratory functions in children with CF of different obstruction severities. Therefore, the aim of this study is to investigate and compare microvascular (endothelium), macrovascular (arterial stiffness) functions in children with CF of different obstruction severities, and to investigate the relationship between micro and macrovascular functions and exercise capacity and respiratory functions in children with CF of different obstruction severities.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is a rare disease with congenital deterioration in mucociliary clearance that causes recurrent or chronic rhinosinusitis, airway infection and bronchiectasis in pediatric age. There are pulmonary genetic disorders associated with inflammation. Children with CF have been shown to have vascular endothelial dysfunction compared to healthy children. Very young children with CF have been reported to have increased arterial stiffness and some decrease in right-left ventricular function. In another study on the subject, it was found that stiffness of the great arteries increased in children with CF; The change in arterial compliancy has been shown to be significant in childhood. The increase in arterial stiffness is associated with systemic inflammation, regardless of blood pressure or diabetes. Hemodynamic changes have been reported in the presence of systemic inflammation in children with CF. Exercise peak workload in children with CF is known to be associated with endothelial dysfunction. It is not known how exercise capacity is affected by endothelial dysfunction and arterial stiffness in CF patients of varying severity. In the literature, there are no studies comparing endothelial function, arterial stiffness and its effect on exercise capacity and pulmonary functions in CF children; this subject is open to research. The aim of this study was to investigate and compare microvascular (peripheral endothelial), macrovascular (arterial stiffness) functions in children with CF and to investigate the relationship of micro and macrovascular functions with exercise capacity and pulmonary functions in children with CF of different obstruction severities.

ELIGIBILITY:
Inclusion Criteria:

* Being clinically stable
* To be cooperated in evaluations to be made
* Forced expiratory volume in the first second (FEV1)> 40%
* No exacerbation in the past three months
* Regular medication for the past 12 months
* No medication changes for at least three weeks

Exclusion Criteria:

* Cardiovascular disease
* Hypertension
* Diabetes
* Pulmonary hypertension
* Smoking
* Resting oxygen saturation (SpO2) <92%
* Using vasoactive drugs (nitrates, b-blockers, angiotensin-converting enzyme inhibitors, etc.)
* Using oral steroids
* Undergoing lung surgery
* Being a highly orthopedic, neurological disease
* Injury to the lower extremity such as injury, sprain, or fracture in the past six months

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who are diagnosed with Cystic Fibrosis with different obstruction severity at Hacettepe University Faculty of Medicine, Department of Pediatric Chest Diseases and who reffered to the Cardiopulmonary Rehabilitation Unit for Physiotherapy also who are willing to participate in the study will be include in the study.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2023-05-02 (Actual)

PRIMARY OUTCOMES:
Maximal exercise capacity | Maximal exercise test will be performed on the first day
  The maximal exercise test will be performed on an electronically braked bicycle ergometer using the Godfrey protocol. The peak work capacity (Wzirve) measurement will be expressed as a percentage of normal values.
Endothelial dysfunction | Endothelial dysfunction assessment will be performed on the first day
  Endothelial dysfunction will be determined by intercellular adhesion molecule-1 (ICAM-1), vascular cell adhesion molecule-1 (VCAM-1), E-selectin, Vascular endothelial growth factor (VEGF), Endothelin-1 (ET-1). Blood samples will be collected.
Arterial stiffness | Arterial stiffness assessment will be performed on the first day
  Arterial stiffness, oscillometric pulse wave velocity (PWV) (m s - 1) and augmentation index (AI@75) (%) will be evaluated by recorded brachial pulse waves with automatically with the oscillometric device.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Inal-Ince, PhD, Study Director — Hacettepe University; Senem Simsek, MSc, Principal Investigator — Hacettepe University; Elmas Ebru Gunes-Yalcin, PhD, Principal Investigator — Hacettepe University; Murat Timur Budak, PhD, Principal Investigator — Hacettepe University; Nagehan Emiralioglu, PhD, Principal Investigator — Hacettepe University; Aslihan Cakmak, MSc, Principal Investigator — Hacettepe University; Yasemin Kartal, MSc, Principal Investigator — Hacettepe University; Suna Sabuncuoğlu, PhD, Principal Investigator — Hacettepe University; Meltem Akgül Erdal, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)